CLINICAL TRIAL: NCT04663607
Title: Randomized Controlled Trial Using Mobile Strategy to Reduce the Risk of Recurrent Preterm Birth
Brief Title: Mobile Strategy to Reduce the Risk of Recurrent Preterm Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of Pittsburgh Medical Center (Other); Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Jason Wang, PROFESSOR OF PEDIATRICS (GENERAL PEDIATRICS) AND HEALTH POLICY, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 54976
Record Dates: First submitted 2020-12-06; First posted 2020-12-11 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Participants will receive paper-based health education as part of standard of care
- PretermConnect App (Experimental): Participants will receive health education via a mobile app, PretermConnect
  Interventions: Behavioral: Use of PretermConnect App

INTERVENTIONS:
Behavioral: Use of PretermConnect App — Participants will receive health education via a mobile app, PretermConnect, in addition to the standard of care, and complete additional surveys on the social determinants of health
  Arms: PretermConnect App

SUMMARY:
Preterm births are defined as delivery prior to 37 weeks gestation and account for 35% of infant deaths in the first year of life. Early preterm birth are deliveries prior to 32 weeks gestation and account for more than 70% of neonatal deaths and 36.1% of overall infant mortality. Women who have delivered a preterm infant and who have a short pregnancy interval (time between giving birth and subsequent conception) have an increased risk of preterm birth in subsequent pregnancies. The investigators hope to understand if a mobile health strategy can be used to reduce spontaneous preterm births via improved patient engagement, care coordination, and adherence to recommended care vs a traditional paper-based health strategy.

DETAILED DESCRIPTION:
The investigators hope to learn how to engage pregnant women at risk for preterm births and reduce the incidence of preterm births through this study. The goal of this study is to reduce the risk of recurrent preterm births for the participating mothers and healthy development of their infants. The investigators hope that this study will accomplish the following for the mothers: Utilize technology to strengthen knowledge of healthy behaviors; Improve adherence to both behavioral and medical interventions that specifically aimed at reducing the risk of spontaneous recurrent preterm births; Develop a platform that can capture participant behavior regarding the participant's lifestyle, environment, social factors, and personal health status; Allow participants to be co-creators of content, thus creating a support network. The investigators hope to achieve improvements in the following primary outcome: Inter-pregnancy interval and the following secondary outcomes: postpartum depression, infant-mother bonding and breast milk feeding between the control and the intervention groups. Ultimately, the investigators hope improvements in these outcomes will improve secondary prevention of preterm births and ultimately reduce infant mortality.

Additionally, PretermConnect will monitor mothers on their social circumstances, such as housing and food insecurity, family employment status, and perceived importance of recommended care for the baby's and the participant's own health.

The investigators also want to observe if a mobile-delivered health management approach can be more effective than a traditional paper-based health management plan in reducing the incidence of subsequent preterm births amongst individuals who have already had at least one preterm birth.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with a mobile phone capable of downloading apps from the Apple App Store or Google Play.
2. Participants must consent to the study.
3. Women whose child is in the neonatal intensive care unit/nursery because the infant was born preterm.
4. Women 16-50 years of age
5. Women who can read, write and understand English

Site-specific additional recruitment criteria

1. UPMC Children's Hospital of Pittsburgh: Mothers whose babies have been in the neonatal intensive care unit for more than one month.
2. UPMC Magee-Womens Hospital: Mothers who have had a preterm baby of <36 weeks.

Exclusion Criteria:

1. For this initial study, those who do not have a mobile phone will be excluded. (This exclusion will not affect the inclusion of minorities as minorities Internet use via mobile platforms is equal to or greater than whites; hence we are not excluding minorities, based on the PEW Research Center study (PEW Internet Spring Tracking Survey, April 17-May 19, 2013)).
2. Women who have not previously had a preterm birth will be excluded as we are trying to reduce the risk of recurrent preterm birth.

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Individuals who have recently delivered a preterm infant
Enrollment: 221 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2025-06-22 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Interpregnancy interval | 12-months
  Time interval from most recent birth to next conception

SECONDARY OUTCOMES:
Breastmilk feeding | 12-months
  Number of participants feeding baby breastmilk by bottle or breast
Postpartum depression | 12-months
  Number of participants that screen for postpartum depression
Mother-infant bonding | 12-months
  Score on mother-infant bonding questionnaire (score range is 10-50; higher scores indicate higher level of bonding)

CONTACTS AND LOCATIONS:
Overall Officials: C. Jason Wang, MD, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - UPMC Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No